CLINICAL TRIAL: NCT06827028
Title: Global Survey on Newborns' HOspitalisation and Parental Experiences
Brief Title: Global Survey on Newborns' HOspitalisation and Parental Experiences - the HOPE Study
Acronym: HOPE
Status: Not yet recruiting | Type: Observational
Sponsor: Global Foundation for the Care of Newborn Infants (Other)
Responsible Party: Principal Investigator, Luc Zimmermann, Professor, Global Foundation for the Care of Newborn Infants
Other Study IDs: METC 2024-0411
Record Dates: First submitted 2024-12-17; First posted 2025-02-14 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Infant, Premature; Infant, Low Birth Weight; Parents; Life Change Events; Needs Assessment; Anxiety; Fear; Stress, Psychological; Uncertainty; Emotions; Caregiver Burden
Keywords: Parental needs; Infant- and Family-centred developmental care; IFCDC; EFCNI; NICU; Global Parent Survey; Breastfeeding; Breastfeeding support; Politics; Needs Assessment; HRQoL; Parents; Infant, Newborn; Family; Family Support; Family Health; Intensive Care, Neonatal; Patient-Centered Care; Infant Care; Surveys and Questionnaires; Health Care Surveys
MeSH Terms: conditions — Premature Birth; Anxiety Disorders; Stress, Psychological; Caregiver Burden; Breast Feeding | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parents/participants: Study participants are parents of newborns that are receiving or received special/intensive care starting within the first week of life and that are born on 1 January 2023 or thereafter. The cohort consists of persons with different ethnic background in different countries that voluntarily participate in the survey.
  Interventions: Other: N/A, no intervention, participation in survey

INTERVENTIONS:
Other: N/A, no intervention, participation in survey — N/A, no intervention, participation in survey

SUMMARY:
This study aims to explore parents' experiences and emotional burdens related to their newborn's hospital stay using an online survey. Our target population consists of parents of newborns born preterm, with low birthweight, or critically ill. Particularly the presence of infant- and family-centred developmental care (IFCDC) principles as well as support through political framework conditions will be investigated.

DETAILED DESCRIPTION:
Collaboration partners, expert working groups and their roles This project will be carried out in close collaboration with representatives of national parent organisations and professional healthcare societies. The following societies are involved as collaboration partners: ANA (African Neonatal Association), CNN (Canadian Neonatal Network), COINN (Council of International Neonatal Nurses), ESPR (European Society for Paediatric Research), NFI (NIDCAP Federation International), UENPS (Union of European Neonatal and Perinatal Societies), WHO Collaborating Centre for Maternal and Child Health. All collaboration partners delegate one representative that supports the Core Working Group (CWG).

The CWG, with n=27 members, and a Support Group (SG), with n=48 members, both consisting of individual multi-professional experts from all continents working in the field of maternal and newborn health, will be assembled. Both groups support the development of the questionnaire in a two-step approach, translations of the questionnaire, the recruitment of participants, data analysis, data interpretation, and publication and dissemination of results. While the CWG, will be actively involved in the initial development of the draft questionnaire, the SG will be involved for a broader review for the revision and final correction of the questionnaire in a second step.

Development of the Questionnaire For the purpose of the HOPE study, we performed a scoping review (1) to explore the available literature related to this topic and to identify the most relevant topics to be included in the questionnaire.

After this literature research, the questionnaire was drafted considering the already existing and validated EMPATHIC-N and the PICKER questionnaires (2,3), as well as the questionnaire, we previously developed to explore parents' experiences related to challenges during the COVID-19 pandemic regarding the care of their newborns (4,5). In addition, questions related to political, social and infrastructural framework conditions were included.

The online questionnaire includes single, multiple choice answer models and some open-text fields. Besides questions related to participant characteristics such as age, sex, country of location, infant birthweight, duration of hospitalisation, etc., the questionnaire includes questions related to the parents' perception of political, social and infrastructural framework conditions as experienced within their country as well as elements of neonatal care mainly involving aspects of IFCDC such as the use and support of breast/human milk and early breast feeding, skin-to-skin care (kangaroo-mother care), parental presence and involvement in the care, shared decision making, stress and pain control etc. during their hospital stay.

In order to maximise the reach and to prevent the loss of study participants due to time constraints, a multi-stage approach will be used, beginning with 47 high-priority questions (single and multiple answer options), followed by more specific second lower-priority questions (single and multiple answer options) (n=21). This first/second layer approach aims to increase the response rate for the most important questions and to keep the effort for participants with limited time resources to a minimum, while taking advantage of the motivation of participants who are willing to share the full scope of their experiences related to their baby's hospitalisation.

The questionnaire draft will be reviewed by the CGW and after having implemented necessary changes, the updated version will be shared with the larger SG for feedback and review. Both groups will ensure that the questionnaire considers the specific national perspective and that the questions are phrased. All implemented changes and the finally updated version of the questionnaire will be discussed with both groups including the representative from the collaboration partners in digital discussion meetings.

In addition, comprehensive interviews with up to 10 participants resembling the target group will be performed to elucidate other relevant topics that may have not yet been covered and need to be included.

The first questionnaire draft (in English) with included feedback from the interviews and experts and will be pre-tested by a comparable target group to receive qualitative feedback on the questionnaire per se and the phrasing.

After a potential adaptation based on data and information of the pre-testing, the questionnaire will be translated in as many different languages as feasible to overcome the linguistic barrier and facilitate participation for parents worldwide. The CWG and SG will support and review the translations. The translated questionnaire versions will be transferred into the online survey software SurveyMonkey ® and will be distributed via the expert groups, GFCNI's network, GFCNI's newsletter and social media channels via an access link.

ELIGIBILITY:
Inclusion Criteria:

Parent or caregiver of a newborn infant born on January 1, 2023, or thereafter, who received/is receiving special/intensive care starting within the first week of life such as oxygen therapy or other respiratory support, incubator treatment, intravenous infusions, treatment of (suspected) sepsis, pneumonia, necrotising enterocolitis, malformations, jaundice, nutritional/feeding problems, hypoglycemia, etc.

Exclusion Criteria:

* Other family members than parents/(primary) caregivers
* Parents of newborns that did not receive special/intensive care starting within the first week of life
* Parents or caregivers of infants born before 1 January 2023
* Persons with insufficient proficiency of one of the languages of the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parent or caregiver of a newborn infant born on January 1, 2023, or thereafter, who received/is receiving special/intensive care starting within the first week of life such as oxygen therapy or other respiratory support, incubator treatment, intravenous infusions, treatment of (suspected) sepsis, pneumonia, necrotising enterocolitis, malformations, jaundice, nutritional/feeding problems, hypoglycemia, etc.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Infant Family-Centered Developmental Care principles | 01/09/2025 - 31/12/2027
  The implementation of IFCDC principles will be measured as the percentage of infants receiving specific care, such as skin-to-skin contact, receiving breastfeeding support, access of parents/caregivers to the neonate, involvement in daily care procedures etc.

SECONDARY OUTCOMES:
Social/Financial/Political Support (Quantitative) | 01/09/2025 - 31/12/2027
  This section will include approximately 10 questions assessing quantitative data on support received by the mother/parents, such as support to access of care, financial compensation for additional expenses (transportation to the hospital, reimbursement for sleeping facilities), social/political support, such as maternity leave etc. The final outcome still depends on the expert decision.
Social/Financial/Political Support (Qualitative) | 01/09/2025 - 31/12/2027
  Subjective qualitative data on support received by the mother/parents, such as support to access of care, financial compensation for additional expenses, social/political support, such as maternity leave etc. indicated by participants via open text fields.
Participant characteristics | 01/09/2025 - 31/12/2027
  Data on Participant characteristics will be collected (such as marital status, parental education etc., and infant characteristics to analyse the influence of these data on the availability of care according the IFCDC principles and describe the study sample.
Questionnaire pre-testing (quantitative) | 01/09/2025 - 31/12/2027
  Quantitative evaluation data of the pre-testing of the questionnaire related to the understandability of questions, utilisation of lay language, appropriateness of selected questions.
Questionnaire pre-testing (qualitative) | 01/09/2025 - 31/12/2027
  Qualitative evaluation data of the pre-testing of the questionnaire indicated in open text fields.

OTHER OUTCOMES:
Single-Country evaluation of IFCDC implementation | 01/09/2025 - 31/12/2027
  The level IFCDC implementation will be analysed per country. Inter-country comparison will be performed to derive recommendations for action.
Single-Country evaluation on the availability of supportive political measures | 01/09/2025 - 31/12/2027
  The availability of supportive political measures will be analysed per country. Inter-country comparison will be performed to derive recommendations for action.

CONTACTS AND LOCATIONS:
Overall Officials: Silke Mader, Study Chair — Global Foundation for the Care of Newborn Health (GFCNI); Helmut Hummler, M.D., M.B.A., Study Director — Global Foundation for the Care of Newborn Health (GFCNI); Luc Zimmermann, Professor, Principal Investigator — Global Foundation for the Care of Newborn Health (GFCNI)
Locations (1):
- Global Foundation for the Care of Newborn Infants (GFCNI), Munich, Bavaria, Germany

REFERENCES:
- [Background] Kostenzer J, Hoffmann J, von Rosenstiel-Pulver C, Walsh A, Zimmermann LJI, Mader S; COVID-19 Zero Separation Collaborative Group. Neonatal care during the COVID-19 pandemic - a global survey of parents' experiences regarding infant and family-centred developmental care. EClinicalMedicine. 2021 Aug 6;39:101056. doi: 10.1016/j.eclinm.2021.101056. eCollection 2021 Sep. PMID 34401688
- [Background] Kostenzer J, von Rosenstiel-Pulver C, Hoffmann J, Walsh A, Mader S, Zimmermann LJI; COVID-19 Zero Separation Collaborative Group. Parents' experiences regarding neonatal care during the COVID-19 pandemic: country-specific findings of a multinational survey. BMJ Open. 2022 Apr 7;12(4):e056856. doi: 10.1136/bmjopen-2021-056856. PMID 35393317
- [Background] Sakonidou S, Kotzamanis S, Tallett A, Poots AJ, Modi N, Bell D, Gale C. Parents' Experiences of Communication in Neonatal Care (PEC): a neonatal survey refined for real-time parent feedback. Arch Dis Child Fetal Neonatal Ed. 2023 Jul;108(4):416-420. doi: 10.1136/archdischild-2022-324548. Epub 2023 Jan 30. PMID 36717224
- [Background] Gill FJ, Wilson S, Aydon L, Leslie GD, Latour JM. Empowering Parents of Australian Infants and Children in Hospital: Translation, Cultural Adaptation, and Validation of the EMpowerment of PArents in The Intensive Care-30-AUS Questionnaire. Pediatr Crit Care Med. 2017 Nov;18(11):e506-e513. doi: 10.1097/PCC.0000000000001309. PMID 28906423
- [Background] Family-centered care in the NICU in a global setting : Ayse Duezenli : Free Download, Borrow, and Streaming. Available from: https://archive.org/details/osf-registrations-erqf7-v1

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-03): https://cdn.clinicaltrials.gov/large-docs/28/NCT06827028/Prot_SAP_001.pdf